CLINICAL TRIAL: NCT00683774
Title: Determination if Direct Inhibition of Insulin Release With Diazoxide Decreases Renal Clearance of D-Chiroinositol (DCI) and Increases Circulating DCI in Obese Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Insulin and Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCU IRB 4479; 2R01HD035629-09A2 (NIH)
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: PCOS
MeSH Terms: interventions — Diazoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCOS subjects (Experimental): PCOS subjects given diazoxide
  Interventions: Drug: diazoxide
- Normal subjects (Active Comparator): Normal subjects given diazoxide
  Interventions: Drug: diazoxide

INTERVENTIONS:
Drug: diazoxide — 100mg orally three times per day for 10 days

SUMMARY:
Increased insulin levels leads to increased secretion of D-chiro inositol(DCI) from the kidneys in women with PCOS, but not in normal women. This leads to a reduction in circulating DCI and insulin stimulated release of DCI-IPG.To determine if decreasing circulating insulin directly by inhibition of islet insulin release with diazoxide in obese women with PCOS 1)decreases the renal clearance of DCI and 2) increases the circulating concentration of DCI.

ELIGIBILITY:
Inclusion Criteria:

* Obese women with PCOS and normal women aged 18-40,
* PCOS less than 8 periods/year, elevated total or free testosterone, normal thyroid function tests and serum prolactin, exclusion of adrenal hyperplasia
* Normal regular monthly periods, no clinical evidence of androgen excess,
* All Acceptable health on interview, medical history, physical exams and lab tests, signed, witnessed informed consent and ability to comply to study requirements

Exclusion Criteria:

* DM, clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic or malignant disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Nestler, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- General Clinical Research Center, Richmond, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.vcu.edu/pcos

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCOS Subjects | Normal Subjects
Started | 11 | 10
Completed | 8 | 9
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Population: Obese women with and without PCOS between the ages of 18-40 years selected after examination and eligibility screening
Groups:
- Total: Total of all reporting groups
Arm/Group | PCOS Subjects | Normal Subjects | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
BMI (Body Mass Index) [Mean (Full Range); unit: kg/m^2] | 41.0 [32.7 to 49.2] | 38.4 [33.3 to 43.4] | 39.7 [32.7 to 49.2]
Waist-to-hip ratio (WHR) [Mean (Full Range); unit: unitless] | 0.84 [0.81 to 0.88] | 0.78 [0.72 to 0.84] | 0.81 [0.72 to 0.88]
Sex hormone binding globulin (SHBG) (nmol/L) [Mean (Full Range); unit: nmol/L] | 32.1 [23.3 to 44.2] | 45.6 [33.7 to 61.7] | 38.9 [23.3 to 61.7]
Total testosterone (ng/mL) [Mean (Full Range); unit: ng/mL] | 2.2 [1.2 to 3.8] | 1.1 [0.6 to 1.8] | 1.7 [0.6 to 3.8]
Free testosterone (pmol/L) [Mean (Full Range); unit: pmol/L] | 144.3 [73.1 to 285.1] | 57.7 [30.4 to 109.6] | 101 [30.4 to 285.1]
Fasting glucose (mg/dl) [Mean (Full Range); unit: mg/dl] | 85.3 [80.7 to 89.9] | 84.2 [77.9 to 90.5] | 84.8 [77.9 to 90.5]
Fasting insulin (ulU/mL) [Mean (Full Range); unit: ulU/mL] | 9.4 [6.7 to 13.1] | 6.8 [5.0 to 9.4] | 8.1 [5.0 to 13.1]
Area under the curve (AUC) glucose (mg*min/dL) [Mean (Full Range); unit: mg*min/dL] | 16447 [15390 to 17504] | 13168 [12209 to 14127] | 14808 [12209 to 17504]
AUC insulin (mg*min/ml) [Mean (Full Range); unit: mg*min/ml] | 8351 [4788 to 14568] | 5284 [3127 to 8929] | 6818 [3127 to 14568]
Whole Body Insulin Sensitivity Index [Mean (Full Range); unit: units on a scale] | 4.76 [2.40 to 7.11] | 6.90 [4.87 to 8.93] | 5.83 [2.40 to 8.93]
Plasma DCI (nmol/mL) [Mean (Full Range); unit: nmol/mL] | 0.36 [0.18 to 0.72] | 0.33 [0.18 to 0.63] | 0.35 [0.18 to 0.72]
24-h urinary D-chiroinositol (DCI) (nmol/day) [Mean (Full Range); unit: nmol/day] | 1808 [927 to 3527] | 1448 [771 to 2719] | 1628 [771 to 3527]
Urinary clearance (uCl) DCI (ml/min) [Mean (Full Range); unit: ml/min] | 3.46 [1.51 to 7.92] | 3.02 [1.38 to 6.59] | 3.24 [1.38 to 7.92]
Plasma myo-Inositol (MYO) (nmol/mL) [Mean (Full Range); unit: nmol/mL] | 19.7 [15.9 to 23.4] | 23.1 [18.9 to 27.3] | 21.4 [15.9 to 27.3]
24-h urinary MYO (nmol/day) [Mean (Full Range); unit: nmol/day] | 52866 [32681 to 85519] | 78909 [50140 to 124184] | 65888 [32681 to 124184]
uCI MYO (ml/min) [Mean (Full Range); unit: ml/min] | 1.91 [1.30 to 2.81] | 2.43 [1.69 to 3.49] | 2.17 [1.30 to 3.49]

OUTCOME MEASURES:

1. Primary Outcome: Renal Clearance of D-chiroinositol (DCI) at 12 Days
Description: Following inhibition of insulin release using diazoxide, measured renal clearance of D-chiro inositol (DCI) via urinary Chiro-inositol dci assay
Time Frame: 12 days
Measure: Mean (Full Range); unit: ml/min
Arm/Group | PCOS Subjects | Normal Subjects
Number analyzed (Participants) | 8 | 9
ml/min | 4.75 [2.25 to 10.01] | 5.16 [2.55 to 10.42]

2. Primary Outcome: Level of Circulating D-chiro Inositol (DCI)
Description: Measured circulating concentration of plasma DCI following inhibition of insulin release using diazoxide
Time Frame: 12 days
Measure: Mean (Full Range); unit: nmol/mL
Arm/Group | PCOS Subjects | Normal Subjects
Number analyzed (Participants) | 8 | 9
nmol/mL | 0.27 [0.12 to 0.57] | 0.27 [0.13 to 0.56]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PCOS Subjects | Normal Subjects
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No